CLINICAL TRIAL: NCT06872021
Title: Early Intra-aortic Balloon Pump Use After Venoarterial Extracorporeal Membrane Oxygenation: The EASE-ECMO Randomized Clinical Trial
Brief Title: Early Intra-aortic Balloon Pump Use After Venoarterial Extracorporeal Membrane Oxygenation
Acronym: EASE-ECMO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS2025197
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: ECMO
Keywords: ECMO; IABP; LV unloading

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECMO+IABP group (Experimental): Patients receive IABP for left ventricular unloading within 6 hours after VA-ECMO initiation.
  Interventions: Other: Early IABP use
- ECMO group (Active Comparator): Patients do not receive mechanical unloading within 6 hours after VA-ECMO initiation.
  Interventions: Other: Conventional approach

INTERVENTIONS:
Other: Early IABP use — Patients receive IABP for left ventricular unloading within 6 hours after VA-ECMO initiation.
  Arms: ECMO+IABP group
Other: Conventional approach — Patients do not receive mechanical unloading within 6 hours after VA-ECMO initiation.
  Arms: ECMO group

SUMMARY:
The goal of this multicenter, randomized trial is to compare early early left ventricular unloading by Intra-aortic Balloon Pump (IABP) versus conventional approach in patients with cardiogenic shock (CS) undergoing venoarterial extracorporeal membrane oxygenation (VA-ECMO). The main question it aims to answer is :

• If left ventricular unloading by IABP as compared with the conventional approach will improve the outcomes in patients undergoing VA-ECMO.

DETAILED DESCRIPTION:
The role of IABP combined with VA-ECMO in patients with CS remains unclear. Therefore, investigators will conduct a prospective randomized clinical trial to explore the effect of early IABP use for LV unloading after VA-ECMO on outcomes in patients with CS. Investigators will randomly assign 358 patients receiving peripheral VA-ECMO to the ECMO+IABP group (n=179) or the ECMO group (n=179). The primary end point was the 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥18
2. Cardiogenic shock(defined as a systolic blood pressure of less than 90 mm Hg for more than 30 minutes or the initiation of catecholamines to maintain a systolic pressure of more than 90 mm Hg, an arterial lactate level of more than 3 mmol per liter, and signs of impaired organ perfusion)
3. Successful implantation of VA-ECMO
4. Informed consent

Exclusion Criteria:

1. Presence of moderate to severe aortic insufficiency or aortic dissection
2. Severe peripheral vascular disease
3. Post-cardiotomy cardiogenic shock(non-CABG procedure) or bridging to cardiac procedure.
4. VA-ECMO for definite non-cardiac causes
5. Extracorporeal cardiopulmonary resuscitation
6. Implantation of IABP or IMPELLA before VA-ECMO
7. Severe bleeding
8. Terminal malignancy
9. Irreversible neurologic injury
10. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days

SECONDARY OUTCOMES:
weaning from VA-ECMO | 30 days
Rate of advanced mechanical unloading | 30 days
Left Ventricular Function of survivors | 30 days
In-hospital Mortality | 30 days
Day of Mechanical Circulatory Support Device Weaning | 30 days
Rate of pulmonary congestion on chest X-ray | 30 days
Duration of VA-ECMO | 30 days
Lactate clearance rate at 12 and 24 hours | 30 days
Relative decrease in vasoactive inotropic score(VIS) at 12 and 24 hours | 30 days
  Vasoactive inotropic score (VIS), in µg/kg/min, was calculated as follows: dopamine + dobutamine + 100 epinephrine + 100 norepinephrine + 15×milrinone. Higher VIS predict worse outome.
Reduction in Myocardial Injury Biomarkers (cTnI/cTnT) | 30 days
Reduction in N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) | 30 days
Rate of CRRT | 30 days
Rate of ventricular arrhythmia | 30 days
Rate of stroke | 30 days
Rate of bleeding | 30 days
  BARC type III or V
Rate of limb ischemia | 30 days
  ECMO side/ IABP side
Duration of mechanical ventilation | 30 days
Rate of infection | 30 days
  With or without culture result
ICU length of stay | 30 days
Hospital length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Hou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No